CLINICAL TRIAL: NCT00874042
Title: A Phase 1 Dose Escalation Study of ARQ 197 Administered in Combination With Gemcitabine in Adult Patients With Advanced Solid Tumors
Brief Title: Dose Escalation Study of ARQ 197 in Combination With Gemcitabine in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-117
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Solid Tumors
Keywords: dose escalation; safety; tolerability; tumor; PK
MeSH Terms: conditions — Neoplasms | interventions — Therapeutics; ARQ 197; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ 197 in combination with gemcitabine (Experimental)
  Interventions: Drug: Treatment with ARQ 197 in combination with gemcitabine

INTERVENTIONS:
Drug: Treatment with ARQ 197 in combination with gemcitabine — Enrollment of an initial cohort of 3 or 6 patients will follow the traditional "3 + 3" dose escalation scheme. These patients will be treated with ARQ 197 and gemcitabine. ARQ 197 will be administered by mouth BID continuously. Gemcitabine will be administered by intravenous infusion over 30 minutes once weekly for 3 consecutive weeks followed by a week of rest.

SUMMARY:
This is an open-label, dose-escalation/de-escalation study of ARQ 197 administered orally in combination with gemcitabine. The study is designed to determine the safety, tolerability and maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of ARQ 197 when administered in combination with gemcitabine to patients with advanced solid tumors.

DETAILED DESCRIPTION:
Enrollment of an initial cohort of 3 or 6 patients will follow the traditional "3 + 3" dose escalation scheme. These patients will be treated with ARQ 197 and gemcitabine. ARQ 197 will be administered by mouth BID continuously. Gemcitabine will be administered by intravenous infusion over 30 minutes once weekly for 3 consecutive weeks followed by a week of rest. The dosing schedules of ARQ 197 and gemcitabine will be as described below.

ARQ 197 will be administered per the following cohorts, starting from week 1 of treatment.

Cohort------ARQ 197 (mg BID)

0-----------120, continuously

1-----------240, continuously

A-----------120 (repeated treatments of 2 weeks followed by a 1 week pause)

B-----------240 (repeated treatments of 2 weeks followed by a 1 week pause)

C-----------360 (repeated treatments of 2 weeks followed by a 1 week pause)

D-----------360 (repeated treatments of 3 weeks followed by a 1 week pause)

E-----------360, continuously

In case of DLT, intermediate dosing cohorts will be explored, administering ARQ 197 for 5 days instead of 7 during the weeks of ARQ 197 administration.

For cohorts 0 and 1, gemcitabine is administered at the dose of 1000mg/sqm from week 1 of treatment, 4 weeks in a row for the first month, then for 3 consecutive weeks followed by a week of pause. For all other cohorts, gemcitabine will be administered starting from week 2 of treatment at the dose of 1000mg/sqm, for 3 consecutive weeks followed by a week of pause.

Additional treatment cohorts may be enrolled to explore intermediate, higher or lower doses of ARQ 197, as indicated by the tolerability, safety profile, and pharmacokinetic (PK) profile.

Once a safe and recommended dose level is determined, an Expanded Cohort of up to 60 patients with non-resectable cholangiocarcinoma (10 patients), breast carcinoma (10 patients), ovarian carcinoma (10 patients), endometrial carcinoma and carcinoma of the cervix (10 patients in total, at least five with endometrial carcinoma). Each group of 10 patients may enroll up to three patients who received at least 5-week gemcitabine treatment. The cohort will also include up to 20 patients with pancreatic carcinoma (up to five out of 20 patients may have received at least 5-week gemcitabine treatment).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent granted prior to initiation of any study-specific screening procedures, given with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* 18 year of age or older
* Histologically or cytologically confirmed locally advanced, inoperable or metastatic primary solid tumors
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5 x ULN with metastatic liver disease
* Hemoglobin ≥ 10 g/dl (or ≥ 9 g/dl for expanded cohort)
* Total bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug
* Male and female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received

Exclusion Criteria:

* Other cancer within the last three years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin
* Previous anti-cancer chemotherapy, radiotherapy, major surgery, immunotherapy or investigational agents within 4 weeks prior to the first day of study defined treatment
* History of cardiac disease: congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD); previously diagnosed bradycardia or other cardiac arrhythmia defined as ≥ Grade 2 according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) (version 3.0), or uncontrolled hypertension; myocardial infarction occurred within 6 months prior to study entry (myocardial infarction occurred > 6 months prior to study entry is permitted)
* Active clinically serious infections defined as ≥ Grade 2 according to NCI CTCAE, version 3.0
* Substance abuse, medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her protocol compliance
* Known human immunodeficiency virus (HIV) infection
* Pregnancy or breast-feeding
* Inability to swallow oral medications
* Significant gastrointestinal disorder, in the opinion of the Investigator, could interfere with the absorption of ARQ 197 and/or gemcitabine (e.g. significant, uncontrolled inflammatory bowel disease or extensive small bowel resection)
* Central nervous system metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability and maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of ARQ 197 when administered in combination with gemcitabine. | Patients will remain on study until unacceptable toxicity, disease progression (clinical or radiological) or another discontinuation criterion is met.

SECONDARY OUTCOMES:
To determine the pharmacokinetic profiles of ARQ 197, gemcitabine and dFdU inactive metabolite of gemcitabine when administered in combination.
To assess the preliminary anti-tumor activity of ARQ 197 when administered in combination with gemcitabine. | Patients will remain on study until unacceptable toxicity, disease progression (clinical or radiological) or another discontinuation criterion is met.
To evaluate dynamic changes of hepatocyte growth factor (HGF), vascular endothelial growth factor (VEGF), and soluble c-Met in patients' peripheral blood that are associated with treatment of ARQ 197 plus gemcitabine. | Patients will remain on study until unacceptable toxicity, disease progression (clinical or radiological) or another discontinuation criterion is met.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Atlanta, Georgia
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Houston, Texas

REFERENCES:
- [Derived] Pant S, Saleh M, Bendell J, Infante JR, Jones S, Kurkjian CD, Moore KM, Kazakin J, Abbadessa G, Wang Y, Chen Y, Schwartz B, Camacho LH. A phase I dose escalation study of oral c-MET inhibitor tivantinib (ARQ 197) in combination with gemcitabine in patients with solid tumors. Ann Oncol. 2014 Jul;25(7):1416-1421. doi: 10.1093/annonc/mdu157. Epub 2014 Apr 15. PMID 24737778